CLINICAL TRIAL: NCT01739777
Title: Phase 1 Randomized-Double Blind Clinical Trial of Intravenous Infusion of Umbilical Cord Mesenchymal Stem Cells Transplantation in Heart Failure on Patients With Cardiopathy in Dilated Stage, of Different Etiology
Brief Title: Randomized Clinical Trial of Intravenous Infusion Umbilical Cord Mesenchymal Stem Cells on Cardiopathy
Acronym: RIMECARD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Responsible Party: Principal Investigator, Jorge Bartolucci, Medical director of Celular Therapy, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UANDES-C4C; CORFO-11IEI-9766 (Other: Government grants)
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Dilated Cardiomyopathy
Keywords: Heart Failure; Coronary Heart Disease; Adult Stem Cells; Umbilical Progenitor Cells; Umbilical Cord Stem Cells Allogenic; Left Ventricular Function; Intravenous Injection
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure; Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ucMSC (Experimental): Umbilical cord derived mesenchymal are injected intravenously to Patients.
  Interventions: Biological: ucMSC
- Controls (Placebo Comparator): Intravenous placebo solution are administrated to Patients.
  Interventions: Other: Controls

INTERVENTIONS:
Biological: ucMSC — 1 million mesenchymal cells per Kg weight injected intravenously in allogenic AB plasma
  Other Names: Umbilical Cord Mesenchymal Stem Cells
  Arms: ucMSC
Other: Controls — Autologous Serum will administrated as placebo
  Arms: Controls

SUMMARY:
The purpose of this study is to determine the safety and clinical effectiveness of umbilical cord mesenchymal cells transplanted by intravenous infusion in patients with heart failure.

DETAILED DESCRIPTION:
Phase I-II Clinical Trial - Safety and efficacy of umbilical cord derived mesenchymal stem cells (ucMSC) in patients with heart failure Randomized, double blind, controlled prospective study in patients with compensated heart failure in dilated phase.

Thirty patients will be selected, who will undergo a strict 3-month followup of ventricular function before being sequentially randomized into two groups: the first group of 15 patients will receive a sole injection of ucMSC and the remaining 15 patients will comprise the control group.

Every patient will maintain their standard treatment of heart failure, with maximum tolerated dosage without side effects.

The day of infusion will be considered day zero. From that moment, followup will be divided into 0-3, 3-6, and 6-12 months.

Clinical results will be analyzed after completion of 12 months of followup.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic heart failure patients in dilated stages
* Etiologies: dilated cardiomyopathy, chronic hypertensive cardiopathy in dilated stage, chronic coronary cardiopathy in dilated stage
* Ejection fraction ≤ 40%.
* Patients who are stable under optimal medical treatment for a period of at least 3 months prior to randomization

Exclusion Criteria:

* Severe or persistent heart failure
* Recurrent myocardial ischemia
* Uncontrolled ventricular tachycardia
* Malignant disease (life expectancy of less than one year)
* Manifest ventricular asynchrony
* Hematologic disease
* Recent cerebrovascular disease
* Recent acute coronary syndrome
* Serum creatinine >2.26 mg/dL (200 umol/L)
* Atrial fibrillation without heart rate control in the last 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
• Change in global left ventricular ejection fraction | 3, 6, 12 months

SECONDARY OUTCOMES:
• Change in functional capacity measured in O2 consumption | 0, 3, 6, 12 months
• Occurrence of major adverse cardiac event | 12 months
• Change in high sensitivity C-reactive protein (hs CRP) | 0, 3, 6, 12 months
• Reduction in level of B-type natriuretic peptide (BNP) | 0, 3, 6, 12 months

OTHER OUTCOMES:
Measures of anti & pro inflammatory cytokines profile | 0-15-90 days
  The cytokine profile we can determinate is Interleukin 1 Beta(IL-1b),Interleukin 6 (IL-6), soluble receptor TNF (TNFRs), tumor necrosis factor(TNF), Interleukin 10 (IL-10), Transforming Growth Factor beta (TGFb), Interferon-gamma (IFNg),Interleukin 17A (IL-17A),Interleukin-4(IL-4) by multiflex flow cytometer.
Change in quality of life | 0-6-12 months
  Measures by specific questionnaire of quality of life:
  Minnesota Living with Heart Failure Questionnaire (MLHFQ). Kansas, City Cardiomyopathy Questionnaire (KCCQ)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Bartolucci, Dr., Principal Investigator — Universidad de Los Andes
Locations (1):
- Universidad de los Andes, Santiago, Chile

REFERENCES:
- [Background] Hare JM, Traverse JH, Henry TD, Dib N, Strumpf RK, Schulman SP, Gerstenblith G, DeMaria AN, Denktas AE, Gammon RS, Hermiller JB Jr, Reisman MA, Schaer GL, Sherman W. A randomized, double-blind, placebo-controlled, dose-escalation study of intravenous adult human mesenchymal stem cells (prochymal) after acute myocardial infarction. J Am Coll Cardiol. 2009 Dec 8;54(24):2277-86. doi: 10.1016/j.jacc.2009.06.055. PMID 19958962
- [Derived] Bartolucci J, Verdugo FJ, Gonzalez PL, Larrea RE, Abarzua E, Goset C, Rojo P, Palma I, Lamich R, Pedreros PA, Valdivia G, Lopez VM, Nazzal C, Alcayaga-Miranda F, Cuenca J, Brobeck MJ, Patel AN, Figueroa FE, Khoury M. Safety and Efficacy of the Intravenous Infusion of Umbilical Cord Mesenchymal Stem Cells in Patients With Heart Failure: A Phase 1/2 Randomized Controlled Trial (RIMECARD Trial [Randomized Clinical Trial of Intravenous Infusion Umbilical Cord Mesenchymal Stem Cells on Cardiopathy]). Circ Res. 2017 Oct 27;121(10):1192-1204. doi: 10.1161/CIRCRESAHA.117.310712. Epub 2017 Sep 26. PMID 28974553
- See also: Universidad de los Andes. — http://www.uandes.cl/